CLINICAL TRIAL: NCT03917966
Title: The Phase II Trial of SHR-1210 Combined With Preoperative Chemotherapy or Apatinib for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: The Phase II Trial of SHR-1210 Combined With Preoperative Chemotherapy or Apatinib for Locally Advanced ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Feng Wang, Director, The First Affiliated Hospital of Zhengzhou University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-02
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: locally advanced esophageal squamous cell carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210+Docetaxel+nedaplatin (Experimental): SHR-1210+Docetaxel+nedaplatin
  Interventions: Drug: SHR-1210+docetaxel+nedaplatin
- SHR-1210+Apatinib (Experimental): SHR-1210+Apatinib
  Interventions: Drug: SHR-1210+Apatinib

INTERVENTIONS:
Drug: SHR-1210+docetaxel+nedaplatin — neoadjuvant chemotherapy:SHR-1210, 200mg,q2w, a total of 3 times; docetaxel 75mg/m2 ivgtt d1, nedaplatin 75mg/m2 ivgtt d1, q3w, for 2 cycles.The patient was evaluated after 2 cycles of neoadjuvant chemotherapy. The surgery was performed 3-4 weeks after the completion of neoadjuvant chemotherapy.
  Arms: SHR-1210+Docetaxel+nedaplatin
Drug: SHR-1210+Apatinib — SHR-1210, 200 mg, q2w; Apatinib, 250mg, qd; 4 weeks is a cycle, a total of 2 cycles
  Arms: SHR-1210+Apatinib

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of SHR-1210 combined with preoperative chemotherapy or Apatinib for locally advanced esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
In China, the incidence of esophageal cancer has declined in recent years, but the mortality rate has been ranked fourth. Morbidity and mortality were ranked sixth and fourth in all malignancies, respectively. Therefore, esophageal cancer has always been a major malignant tumor that threatens the health of our residents. Investigator designed a single-arm, open-label, phase II trial of SHR-1210 combined with preoperative chemotherapy or Apatinib for locally advanced esophageal squamous cell carcinoma. The purpose of this study is to observe and evaluate the efficacy and safety of SHR-1210 combined with preoperative chemotherapy or Apatinib for locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, both men and women;
2. Histology confirmed as esophageal squamous cell carcinoma;
3. Resectable stage Ⅱ/Ⅲ/Ⅳa（cT2-4aN0-3M0）;
4. ECOG: 0~1;
5. Expected survival period≥12 weeks;
6. The main organs function normally, that is, the following criteria are met:(1)Blood routine examination:a.HB≥90g/L; b.ANC≥1.5×109 / L; c.PLT≥80×109 / L (2)Biochemical examination:a.ALB≥30g / L; b.ALT and AST≤2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN; c.TBIL ≤1.5ULN;d.plasma Cr≤1.5ULN or creatinine clearance (CCr) ≥ 60ml / min;
7. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%);
8. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy test within 7 days prior to study enrollment And must be non-lactating patients; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period;
9. Subjects voluntarily joined the study, signed informed consent, and were well-adhered to follow-up;
10. Can swallow tablets normally.

Exclusion Criteria:

1. Does not meet the above inclusion criteria;
2. Those who are allergic to or sensitive to Docetaxel and nedaplatin;
3. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis,Hyperthyroidism; patients with vitiligo; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
4. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppressive purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used for 2 weeks prior to enrollment;
5. Patients with any severe and/or uncontrolled diseases:Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg); myocardial ischemia or myocardial infarction with grade I or above, arrhythmia (including QT interval ≥480ms) and grade I cardiac insufficiency;
6. Active or uncontrolled serious infections;
7. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 104 copies/ml or 2000 IU/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method);
8. Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0g;
9. Pregnant or lactating women;
10. Patients with other malignancies within 5 years (except for basal cell carcinoma and cervical carcinoma in situ) that have been cured;
11. Patients with a history of psychotropic substance abuse who are unable to quit or have a mental disorder;
12. Patients who have participated in other drug clinical trials within four weeks;
13. At the discretion of the investigator, there are patients with serious concomitant disease that compromises patient safety or affects the patient's completion of the study;
14. The investigator believes that it is not suitable for inclusion;
15. Patients with esophageal squamous cell carcinoma whose primary focus is active bleeding;
16. With active ulcer, unhealed wound or fracture;
17. Suffer from hypertension and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
18. Abnormal coagulation function (INR > 2.0 or prothrombin time (PT) > 16S), bleeding tendency or undergoing thrombolytic or anticoagulant therapy (preventive use of low-dose aspirin and low molecular weight heparin is allowed);
19. Patients with clinically significant bleeding symptoms or definite bleeding tendency within the first three months of randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis, can be reexamined if the stool occult blood is positive in the baseline period. If it is still positive after reexamination, endoscopic examination is required (except those who have accepted endoscopic examination within three months before enrollment and excluded such cases);
20. Arteriovenous thrombosis events occurred within the first 6 months of randomization, such as cerebrovascular accidents (including transient ischemic attack, intracerebral hemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism;
21. Known hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, etc.);
22. Routine urine examination showed that urinary protein was ≥ + + and it was confirmed that the amount of urinary protein in 24 hours was > 1.0 g;
23. Patients with supraclavicular lymph node metastasis; Poor nutritional status, BMI < 18.5 kg / m2; If it is corrected before randomization after symptomatic nutritional support, it can continue to be considered after evaluation by the main investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2023-10-07 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
Major pathological response（MPR） | At time of surgery
  defined as ≤ 10% residual viable tumor at the time of surgical resection, as assessed by central pathology laboratory.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | At time of surgery
  defined as the absence of any viable tumor at the time of surgical resection, as assessed by central and local pathology laboratory
Overall Survival (OS) | up to 2 year
  defined as the time from randomization to death from any cause during the course of the study.
Disease-Free Survival (DFS) | up to 2 year
  Time after R0 resection to disease recurrence or death
Lymph node derating rate | At time of surgery
  Lymph node derating rate
R0 resection rate | At time of surgery
  R0 resection rate

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China